CLINICAL TRIAL: NCT03491605
Title: Study to Surveil and Track the Outcomes of Chronic Latent EBV Infection Based on Healthy Volunteers Undergoing Routine Inspection
Brief Title: Surveillance and Tracking the Outcomes of Chronic Latent EBV Infection
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jianfeng Zhou, Director of Hematology,Tongji Hospital,Tongji Medical College, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Other Study IDs: TJH0002017
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: EBV Infection
Keywords: chronic EBV infection, hemophagocytic lymphohistiocytosis
MeSH Terms: conditions — Epstein-Barr Virus Infections; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. perepheral blood sample of the subjects who have high load peripheral EBV-DNA
  2. tumor tissues of the subjests who progress to hematological malignancies during the follow-up process
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- peripheral EBV-DNA load: subjects with high load (>1×103 copies/ml）of EBV-DNA copies in peripheral blood.
  Interventions: Other: peripheral EBV-DNA load

INTERVENTIONS:
Other: peripheral EBV-DNA load — No intervention

SUMMARY:
Immunocompetent subjects with high load of Epstein-Barr virus DNA (EBV-DNA) in peripheral blood will be enrolled and prospectively followed up to track the natural histories of the chronic high load of EBV virus. The primary goal of this study is to explore the association of peripheral high load of EBV with the hematological malignancies, and second goal is to investigate the genetic mechanisms of immune escape and tumorigenesis of chronic EBV infection.

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) is an oncogenic virus implicated in the pathogenesis of a variety of human hematological malignancies such as lymphomas, hemophagocytic lymphohistiocytosis and chronic active EBV disease. While chronic latent EBV infection（especially carriers with persistent high load of EBV-DNA copy number）is the gray zone between the primary infection and the hematological malignancies, which is rarely concerned. Previous work has prompted the heterogeneities of EBV infection, such as racial heterogeneity, viral load heterogeneity and heterogeneity of infected target cells. It is of great significance to prospectively track the transforming process and elucidate the association of chronic EBV infection and hemophagocytic lymphohistiocytosis. Healthy subjects who was found to have high EBV-DNA load （>1×103 copies/ml）in peripheral blood during the physical examination were enrolled and followed up by telephone or face-to-face interview periodically. The primary outcome is hematological malignancies including Burkitt lymphoma, EBV+ B-cell lymphoproliferative diseases, extranodal NK/T-cell lymphoma of nasal type (ENKL), aggressive NK-cell leukemia (ANKL), classic Hodgkin lymphoma,EBV-associated hemophagocytic lymphohistiocytosis and Chronic active Epstein-Barr virus infection (CAEBV). The Exploratory purpose of this study is to investigate of genetic mechanisms of immune escape and tumorigenesis of EBV infection. Subgroup analysis will performed in subjects with mild high load (>1×103 copies/ml and <1×104 copies/ml) and severe high load (>1×104 copies/ml) of EBV-DNA copies.

ELIGIBILITY:
Inclusion Criteria:

1. immunocompetent subjects who was found to have high EBV-DNA load （>1×103 copies/ml）in peripheral blood during the physical examination
2. Willing to be followed up by telephone or face-to-face interview

Exclusion Criteria:

1. Subjects with defined immunodeficiency
2. Subjects who have taken or are going to take immunosuppressive drugs.
3. Subjects Diagnosed a validated hematopathy
4. Subjects diagnosis as precancerous lesion or malignant tumor and the life expectancy is less than 1 year.
5. psychological illness which does not allow subjects to understand the study and participate following his own free will
6. Pregnant woman
7. no written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of immunocompetent subjects with high load (>1×103 copies/ml) of Epstein-Barr virus DNA (EBV-DNA) in peripheral blood will be enrolled and prospectively followed up to track the natural histories of the chronic latent EBV infection.The subjects were enrolled from healthy examers in Tongji Hospitoal attached to Huazhong University of Science and Techonology. There is no limitation regarding to age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
hematological malignancies | Five years or more if necessary
  including Burkitt lymphoma, EBV+ B-cell lymphoproliferative diseases, extranodal NK/T-cell lymphoma of nasal type (ENKL), aggressive NK-cell leukemia (ANKL), classic Hodgkin lymphoma, and Chronic active Epstein-Barr virus infection (CAEBV).

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Zhou, PhD.and MD., Study Chair — Director of Department of Hematology in Tongji Hospital，HUST
Locations (1):
- Tongji hospital, Tongji medical collage of HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.